CLINICAL TRIAL: NCT05489003
Title: Fatigue, Psychological Comorbidity and Quality of Life Among Patients With Chronic Pancreatitis in China.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: XH20220802
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Chronic Pancreatitis
Keywords: Chronic pancreatitis; Fatigue; Anxiety; Depression; Quality of life
MeSH Terms: conditions — Pancreatitis, Chronic; Fatigue; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with fatigue: Chronic pancreatitis patients with fatigue measured by professional assessment scales.
- Patients without fatigue: Chronic pancreatitis patients without fatigue measured by professional assessment scales.

SUMMARY:
This study will investigate the status of fatigue, psychological comorbidity and quality of life among patients with chronic pancreatitis in China and analyze their influencing factors.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is an inflammatory disease characterized by pancreatic fibrosis. Available studies suggested that the incidence of CP in China was about 13.5 per 100,000 people. Patients with CP often have symptoms of pancreatic endocrine and exocrine insufficiency such as elevated blood sugar, weight loss, muscle loss, combined with complications such as pancreatic duct stones, pancreatic duct stenosis, pancreatic pseudocysts, and have a higher risk of pancreatic cancer, which seriously affects the quality of life of patients.

Psychological comorbidities represented by anxiety and depression were thought to be widespread in CP patients, with available epidemiological studies indicating that the prevalence of anxiety and depression in CP patients in the United States was 36.8% and 46.8%, respectively. In addition, fatigue, as a subjective perception of decreased ability to perform physical and/or intellectual tasks, has also been founded among CP patients.

However, to date, there is a lack of epidemiological studies on fatigue, anxiety, depression and quality of life in Chinese patients with CP. This study will investigate the epidemiological status of fatigue, anxiety, depression, and quality of life in Chinese patients with CP and analyze the factors influencing them.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic pancreatitis

Exclusion Criteria:

* Illiterate
* Having communication difficulties
* Unable to complete the questionnaires
* Having a history of psychiatric disorders
* Recent history of psychotropic and sedative drug use
* Pregnancy
* Rejected participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pancreatitis in China.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of fatigue among patients with CP in China. | Within 1 month after data analysis.
  The level of fatigue in CP patients was measured using the Multidimensional Fatigue Inventory (MFI-20), and the Fatigue Severity Scale (FSS).
The incidence of anxiety among patients with CP in China. | Within 1 month after data analysis.
  The level of anxiety in CP patients is measured using the Hospital Anxiety and Depression Scale (HADS), and the Zung Self-Rating Anxiety Scale (SAS).
The incidence of depression among patients with CP in China. | Within 1 month after data analysis.
  The level of anxiety in CP patients is measured using the Hospital Anxiety and Depression Scale (HADS), and the Zung Self-rating Depression Scale (SDS).
The incidence of quality of life among patients with CP in China. | Within 1 month after data analysis.
  The level of quality of life in CP patients is measured using the European organization for the research and treatment of cancer QOL questionnaire (EORTC-QLQ C-30).

SECONDARY OUTCOMES:
The influencing factors of fatigue among patients with CP in China. | Within 1 month after data analysis.
  Factors included are obtained from the patient's electronic medical record or by asking the patient directly. The content mainly included (1) sociodemographic data: age, gender, education level, income level, marital status, social support level, and patient's life history (smoking and alcohol consumption), etc; (2) clinical data of CP: first symptoms, frequency of abdominal pain, severity of pain, and times of hospitalization for acute pancreatitis, etc; and (3) patient's psychological conditions: the level of anxiety and depression.
The influencing factors of anxiety and depression among patients with CP in China. | Within 1 month after data analysis.
  Factors included are obtained from the patient's electronic medical record or by asking the patient directly. The content mainly included (1) sociodemographic data: age, gender, education level, income level, marital status, social support level, and patient's life history (smoking and alcohol consumption), etc; (2) clinical data of CP: first symptoms, frequency of abdominal pain, severity of pain, and times of hospitalization for acute pancreatitis, etc.
The influencing factors of depression among patients with CP in China. | Within 1 month after data analysis.
  Factors included are obtained from the patient's electronic medical record or by asking the patient directly. The content mainly included (1) sociodemographic data: age, gender, education level, income level, marital status, social support level, and patient's life history (smoking and alcohol consumption), etc; (2) clinical data of CP: first symptoms, frequency of abdominal pain, severity of pain, and times of hospitalization for acute pancreatitis, etc.
The influencing factors of quality of life among patients with CP in China. | Within 1 month after data analysis.
  Factors included are obtained from the patient's electronic medical record or by asking the patient directly. The content mainly included (1) sociodemographic data: age, gender, education level, income level, marital status, social support level, and patient's life history (smoking and alcohol consumption), etc; (2) clinical data of CP: first symptoms, frequency of abdominal pain, severity of pain, and times of hospitalization for acute pancreatitis, etc; and (3) patient's psychological conditions: the level of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Hao Hu, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No